CLINICAL TRIAL: NCT06026917
Title: A Single-Arm, Open-Label, Exploratory Mechanistic Validation (PoM) Clinical Trial of Toludesvenlafaxine Hydrochloride Extended-Release Tablets Assessing Dopamine Transporter Occupancy in the Patients With Depression Brain Using 11C-CFT Positron Emission Tomography (PET)
Brief Title: Assessing Dopamine Transporter Occupancy in the Patients With Depression Brain With Toludesvenlafaxine Hydrochloride Extended-Release Tablets Using 11C-CFT Positron Emission Tomography (PET)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Yantai University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMHC-235
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toludesvenlafaxine hydrochloride sustained-release tablets (Experimental): 40 mg/tablet, 80mg/tablet, 40 mg~160mg each time, once a day, for 42 days
  Interventions: Drug: Toludesvenlafaxine hydrochloride sustained-release tablets

INTERVENTIONS:
Drug: Toludesvenlafaxine hydrochloride sustained-release tablets — D1~D6, 40mg/ tablet, 1 tablet per time, once a day, D7~D10, 80mg/ tablet, 1 tablet per time, once a day, D11~D42, 80mg/ tablet, 2 tablets per time, once a day. For subjects who cannot tolerate 160mg, the dose may be reduced to 80mg/ dose once daily. After the number of subjects receiving 160mg/ dose reached 6, the remaining subjects received D11~D42, 80mg/ tablet, one tablet each time, once a day.

SUMMARY:
This study was a single-arm, open-label clinical study to assess dopamine transporter occupancy in the brain of patients with depression using 11C-CFT positron emission tomography (PET).

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients aged 18 years and older;
* Meet DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition) diagnostic criteria for depression (296.2/296.3), and not accompanied by psychotic features;
* A Montgomery - Asberg Depression Rating Scale (MADRS) total score ≥ 26 at screening;
* Anhedonia scale score < 28.5 at screening;
* Subjects and their partners take effective non-drug contraceptive measures (such as abstinence and condom with intravaginal spermicide) throughout the study and within 6 months after the end of the study, and have no sperm donation plan;
* The subject is willing to participate in the trial and sign the informed consent form and is able to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

* Known to have a history of allergy to any component of the investigational drug or similar drugs, or allergic constitution (defined as allergy to two or more drugs or food) and the investigator determines that it is not appropriate to participate in the trial;
* Significant suicide attempt or behavior, MADRS scale item 10 (suicidal ideation) score ≥ 4 points;
* Pregnant or lactating women, recently planned pregnancy;
* Those who meet DSM-5 diagnosis of schizophrenia spectrum or other psychoses, bipolar or related disorders, obsessive-compulsive and related disorders, traumatic and stress-related disorders, dissociative disorders, anorexia nervosa or bulimia, personality disorders, substance-related or alcohol use disorders (except nicotine or caffeine);
* Patients with depression secondary to other mental or physical diseases or with a past medical history or family history of movement disorders (such as Parkinson's disease);
* Receipt of any contrast agent or radiopharmaceutical within 48 hours before the application of the trial drug, or planned application of contrast agent within 24 hours after the administration of the trial drug;
* Contraindications to PET or MRI (magnetic resonance imaging) (including claustrophobia, alcohol allergy, cardiac pacemaker and neurostimulator in the body, metal foreign body or tracer component allergy, etc.); in the past 10 years,Major occupational exposure to ionizing radiation (e.g., more than 50 nanovolts/year) or exposure to radioactive substances or ionizing radiation for therapeutic or research purposes;
* Patients who stopped antidepressant drugs for less than 7 half-lives (at least 2 weeks for monoamine oxidase inhibitors and at least 1 month for fluoxetine) before entering the group;
* History of gastrointestinal disease known to interfere with drug absorption or excretion or history of surgery known to interfere with drug absorption or excretion;
* History of increased intraocular pressure or narrow glaucoma;
* Total bilirubin (TBIL) value 1.5 times higher than the upper limit of normal, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 3 times higher than the upper limit of normal, thyroid stimulating hormone (TSH) higher than the normal range or glomerular filtration rate (GFR) ≤ 70 mL/min at screening or baseline;
* Patients with serious unstable cardiovascular disease, liver disease, kidney disease, blood disease, endocrine disease, central nervous system and other physical diseases or medical history, or the subjects are not suitable for the study judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Dopamine Transporters Occupancy in the Basal Ganglia（Positron emission tomography with 11C-CFT） was determine by SUVr of the Basal Ganglia DAT. | from baseline to day 14 and 42

SECONDARY OUTCOMES:
Changes in the total score of 10 items on the Montgomery-Asperger's Depression Scale (MADRS) from baseline | from baseline to day 42
Changes in the Scores anhedonia | from baseline to day 42
Incidence Rate of Adverse event | from baseline to day 42

CONTACTS AND LOCATIONS:
Overall Officials: YIFENG SHEN, MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No